CLINICAL TRIAL: NCT03875911
Title: A Prospective Randomized Clinical Trial Comparing Three Delivery Methods of Mitomycin-C for Trabeculectomy Surgery: Preoperative Subconjunctival Injection, Intraoperative Subconjunctival Injection, and Topical Application (Conventional Use) During Trabeculectomy Surgery
Brief Title: Comparing Preoperative Injection of Mitomycin-C vs. Intraoperative Injection of Mitomycin-C vs. Topical Application of Mitomycin-C (Conventional Use) in Trabeculectomy
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Problems unique to COVID-19, incomplete data due to a high rate of dropout to minimize non-essential appointments and difficult subject recruitment
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Joseph Caprioli, Distinguished Professor of Ophthalmology and David May II Chair in Ophthalmology, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-000432
Record Dates: First submitted 2019-03-13; First posted 2019-03-15 (Actual); Results first posted 2024-01-05 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Glaucoma Open-Angle Primary; Glaucoma; Open Angle Glaucoma; Glaucoma, Open-Angle
Keywords: Trabeculectomy; Mitomycin-C; Glaucoma
MeSH Terms: conditions — Glaucoma, Open-Angle; Glaucoma | interventions — Mitomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Preoperative Subconjunctival injection of MMC (Active Comparator): Subconjunctival injection of 0.1 ml of Mitomycin-C 0.002% at the site of future trabeculectomy surgery (2 - 4 weeks preoperatively).
  Interventions: Drug: Mitomycin C
- Intraoperative subconjunctival injection of MMC (Active Comparator): Intraoperative subjconjunctival injection of 0.1 mL of Mitomycin-C 0.01% (0.1mg/mL) to the site of trabeculectomy
  Interventions: Drug: Mitomycin C
- Intraoperative topical application of MMC (Active Comparator): Topical application of Mitomycin-C intraoperatively by applying a sponge soaked in 1mL of Mitomycin-C 0.02 mg/mL for 1 minute to the site of trabeculectomy
  Interventions: Drug: Mitomycin C

INTERVENTIONS:
Drug: Mitomycin C — Three delivery methods of Mitomycin-C in Trabeculectomy

SUMMARY:
In this Pilot explorative study, the investigators are going to estimate and compare the outcomes of three different delivery methods of MMC for Trabeculectomy: a subconjunctival injection of MMC 0.002% at the site of future Trabeculectomy two to four weeks before the surgery, a subconjunctival injection of MMC 0.01% intraoperatively and topical sponge applied MMC 0.02% intraoperatively (typical use) in patients with Primary Open Angle Glaucoma who did not have any filtering surgeries before.

After obtaining informed consent from the patients, the patients are randomly divided into three groups via a block randomization method: Group A receives 0.1 mL MMC 0.002 % (0.1mL MMC 0.02mg/mL) subconjunctival injection preoperatively in superior conjunctiva at the site of future Trabeculectomy surgery. Group B receives 0.1mL MMC 0.01% subconjunctival injection intraoperatively at the site of Trabeculectomy and Group C receives conventional sponge delivery of MMC 0.02% intraoperatively. To avoid observer bias during postoperative evaluation of results, IOP staff obtaining measurements of IOP will be masked to the randomization allocation.

All groups undergo conventional Trabeculectomy surgery (fornix-based) as scheduled, and the same routine follow up and post-op regimen will be scheduled for all three groups. Patients are routinely visited in the clinic at first day postoperatively, one week (+/-2 days), one month (+/-1 week), three months (+/-2 weeks), six months (+/-3 weeks) and finally at one year (+/-(4 weeks)). In each of these visits we will be assessing: Visual acuity, intraocular pressure, number and type of glaucoma medication, slit lamp examination of the anterior segment and fundus examination.

DETAILED DESCRIPTION:
Purpose:

To obtain estimates of the effect on intraocular pressure and side effects of three delivery methods of Mitomycin C (MMC) compared among each other: preoperative subconjunctival injection of 0.1 mL MMC 0.002%, subconjunctival injection of 0.1 mL MMC 0.01% intraoperatively, and conventional sponge applied MMC (0.02%) during trabeculectomy surgery in patients with Primary Open Angle Glaucoma who did not have any filtering surgeries before.

Objective:

To obtain estimates for intraocular pressure reduction among three delivery methods of MMC compared among each other: preoperative subconjunctival injection, intraoperative subconjunctival injection, and intraoperative topical use during trabeculectomy surgery, and to report any associated adverse effects.

Null hypothesis:

There is no use of hypothesis testing in this pilot study.

Alternative hypothesis:

There is no use of hypothesis testing in this pilot study.

The effect and safety of MMC subconjunctival injection either preoperatively or intraoperatively has been previously investigated in Pterygium surgery (Khakshoor H, Razavi ME, Daneshvar R, Shakeri MT, Ghate MF, Ghooshkhanehi H. Am J Ophthalmol. 2010 Aug;150(2):193-8. Preoperative subpterygeal injection vs intraoperative mitomycin C for pterygium removal: comparison of results and complications).

Previous studies comparing effectiveness of subconjunctival injection of MMC vs sponge-applied MMC have shown inconsistent results. In one retrospective study, Mitomycin-C applied by injection resulted in significantly lower IOP, and the need for fewer glaucoma medications, however description of methods is incomplete. (Lim MC. A comparison of trabeculectomy surgery outcomes with mitomycin-C applied by intra-Tenon injection versus sponge method. American Glaucoma Society 23rd Annual Meeting; 2013, San Francisco, CA). One retrospective study showed similar efficacy and safety of intraoperative MMC injection compare to sponge application in trabeculectomy surgery with overall lower IOP in the injection group and main advantages being a large surface area of exposure and a predictable dose of deliver when the injection was performed. No difference in postoperative complications between groups was observed. A small sample size (30) in each group might prevent finding statistical significant results. (Khouri AS, Huang G, Huang LY. Intraoperative Injection vs Sponge-applied Mitomycin C during Trabeculectomy: One-year Study. J Curr Glaucoma Pract 2017;11(3):101-106). A previous case report on preoperative administration of MMC for Trabeculectomy showed reduction of IOP with short follow-up (6 months) Hung PT, Lin LL, Hsieh JW, Wang TH. Preoperative mitomycin-C subconjunctival injection and glaucoma filtering surgery. J Ocul Pharmacol Ther. 1995;11(3):233-241.

One RCT with a follow-up of 3 years compared outcomes of intraoperative injection versus sponge-applied MMC and no significant difference in IOP was found however a more favorable bleb morphology was found in the injection group which is correlated with better function and long-term success of Trabeculectomy ( Esfandiari, Hamed et al. Treatment Outcomes of Mitomycin C-Augmented Trabeculectomy, Sub-Tenon Injection versus Soaked Sponges, after 3 Years of Follow-up Ophthalmology Glaucoma , Volume 1 , Issue 1 , 66 - 74)

In this study the comparison will be the timing and route of delivery of MMC in all three groups, having found inconsistent reports in the literature and very scarce data on the effect of preoperative subconjunctival MMC the investigators would like to further explore in this pilot study the effect of subconjunctival injection on IOP reduction for trabeculectomy at preoperative and intraoperative phases. Since there is no group receiving placebo, the inclusion of a sham injection will not affect the outcomes compared to GROUP C and could increase preoperative risks to patients. The same methodology has been applied in two previous randomized controlled trials. (Pakravan M, Esfandiari H, Yazdani S, et al. Mitomycin C-augmented trabeculectomy: subtenon injection versus soaked sponges: a randomized clinical trial Br J Ophthalmol 2017;101:1275-1280 and Khan F, Niazi S, Awais M et all. Effectiveness of Preoperative Subconjunctival Injection of Mitomycin-C in Primary Pterygium Surgery Journal of the College of Physicians and Surgeons Pakistan 2017, Vol. 27 (2): 88-91)

Glaucoma patients who need glaucoma surgery, such as trabeculectomy, have ongoing damages that cannot be managed only with medication such as drops, and pressure reduction is absolutely crucial in preserving visual function in these patients, hence any possible action that can add to this reduction is valuable.

On the other hand, there are several risks associated with the topical applied MMC usage at the time of surgery mainly due to the inability to precisely quantify the amount of MMC delivered by the sponge application which was shown to be far less with the injection of MMC by delivering a predicted volume either at surgery or before the surgery which are mentioned in the first two paper references.

The selected concentrations for the MMC injection are based on pharmacological studies performed on ocular tissue in which the concentration achieved after subconjunctival injection was established.

STUDY DESIGN This is a multicenter, randomized, controlled pilot study with a main objective of obtaining estimates of differences in IOP reduction among three methods of delivery of mitomycin C for use in trabeculectomy surgery.

The injectors and patients are unmasked in this study while the evaluators are masked.

This study will be performed at the Glaucoma Division of Stein Eye Institute-UCLA Los Angeles, CA.

METHODS

Patients who met inclusion criteria and had signed an informed consent will then be randomized into three groups as follows:

* Group A: Patients will receive a subconjunctival injection of 0.1mL MMC 0.02mg/mL which corresponds to 0.002% (a tenth of the concentration of conventional topical MMC use) at the site of future trabeculectomy surgery two to four weeks in advance. A follow-up phone call 1 week after the MMC injection will assess any side effects of the procedure. If side effects are reported by the patient an appointment will be schedule for a follow up in-office visit and appropriate treatment will be delivered. On the day of conventional trabeculectomy no MMC will be injected. Follow-up will be scheduled for one year.
* Group B: On the day of conventional trabeculectomy patients will receive a subconjunctival injection intraoperatively of 0.1 mL MMC 0.1mg/mL which corresponds to 0.01% (half the concentration of conventional topical MMC use) at the site of trabeculectomy. Surgeon will irrigate the surface of the eye after MMC injection to remove any MMC that might have leaked out. Follow-up will be scheduled for one year.
* Group C: On the day of conventional trabeculectomy patients will receive MMC by applying a sponge soaked in 1mL of MMC 0.2 mg/mL (0.02%) for 1 minute to the site of trabeculectomy surgery followed by irrigation. MMC is standard of care for trabeculectomy surgery at UCLA. This differs from the proposed research because the MMC will be administered as an injection either two to four weeks before the surgery in Group A or intraoperatively in Group B rather than the usual topical administration on the day of surgery (Group C). Follow-up will be scheduled for one year.

The concentration of MMC in each group were chosen according to the delivery method and the timing of exposition of the tissue to the MMC in order to prevent complications from overdose. Based on experimental studies on ocular tissues that evaluated the final amount of MMC delivered to scleral tissue and finding a similar result when using subconjunctival injection of 0.02% with immediate irrigation and 0.002% without irrigation, the investigators chose the latter for group A. Few studies evaluated MMC subconjunctival injection one month before pterygium surgery using 0.02% and 0.015% with a follow-up of 3 years establishing safety of this approach. For group B the investigators chose a similar methodology of a previous RCT comparing subconjunctival injection versus topical administration of MMC for trabeculectomy that used a reduced concentration of 0.01%.

Data collection will be as follows: At preoperative visit, postoperative day one, one week (+/- 2 days), one month (+/- 1 week), three months (+/- 2 weeks), six months (+/- 3 weeks) and one year (+/- 4 weeks). The data will be recorded in the REDCap (Research Electronic Data Capture) software which has free access and allows for easy recording and uploading of imaging (VF, Optic nerve OCT, AS-OCT and bleb photography) for future analysis.

In each of these visits, the following data will be collected: Visual acuity, intraocular pressure, number and type of glaucoma medication, slit lamp examination of the anterior segment, fundus examination and adverse events if present. Visual field and optic nerve OCT will also be included in the preoperative evaluation and at 12 months postoperatively.

For better assessment of the bleb morphology, the investigators will include a clinical grade system, slit lamp photography, and AS-OCT [Anterior segment module of Spectralis OCT device (Heidelberg Engineering, Inc., Heidelberg, Germany)] of the bleb.

For the clinical description of the bleb and a more standardized comparison of the morphological changes over time, the investigators included at every postoperative visit the description of the bleb using the Moorfields Bleb Grading System (MBGS) which captures more morphological features and regional vascularity compared to other systems. (Wells AP, Ashraff N, HalL RC et all Comparison of Two Clinical Bleb Grading Systems Ophthalmology 2006;113:77-83).

The bleb photography will be included at the Month 3 and Month 12 postoperative visits and AS-OCT at 1,3,6 and 12 Month follow-ups. The inclusion of AS-OCT allows for evaluation of the internal structure of the bleb that has been shown to have prognostic implications for outcomes of surgery. Kokubun T, Tsuda S, Kunikata H et all. Anterior-Segment Optical Coherence Tomography for Predicting Postoperative Outcomes After Trabeculectomy, Current Eye Research, DOI: 10.1080/02713683.2018.1446535

Block randomization:

To ensure the balance of sample size between three treatment groups, block randomization is used for treatment assignment. Specifically, each block consists of 6 patients, including 2 patients in each of three treatment groups, and all possible permutations of a sequence of treatment assignment for these 6 patients are generated, such as AABBCC, ABCABC, etc. A random number is then generated to select a block of treatment assignment for 6 patients among all possible blocks, and a sequence of such random blocks will form the sequence of treatment assignment for all patients after their enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Age: 20 - 85 years
* Willingness to participate in the study by signing informed consent
* Primary open angle glaucoma (including pigmentary glaucoma and pseudoexfoliation glaucoma) indicated with open angles upon previous gonioscopy and demonstrative optic nerve and visual field damage
* Trabeculectomy needed as treatment as determined by the care provider

Exclusion Criteria:

* Patient unwilling or unable to give informed consent, unwilling to accept randomization, or unable to return for scheduled study visits throughout the duration of the study (1 year)
* Any secondary cause of glaucoma, or angle closure shown on gonioscopy
* Any ocular or neurological problems with optic nerve or visual field defect (ie. retinal disease, post trauma, corneal scar) that may confound the interpretation of glaucoma such as visual field or optic nerve interpretation
* Pregnant women, nursing women, and/or anyone with a history of allergy to MMC

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2019-03-30 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Doheny Eye Center UCLA (Arcadia), Arcadia, California
  - Doheny Eye Center UCLA (Fountain Valley), Fountain Valley, California
  - Stein Eye Institute - UCLA (Westwood), Los Angeles, California
  - Doheny Eye Center UCLA (Pasadena), Pasadena, California

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Eyes
Groups:
- Group A - Pre-operative Injection: Recieved a pre-operative injection of mitomycin-C prior to trabeculectomy
- Group B - Intra-operative Injection: Recieved an intra-operative injection of mitomycin-C
- Group C - Control: Recieved standard of care - topical application of mitomycin-C
Period: Overall Study
Arm/Group | Group A - Pre-operative Injection | Group B - Intra-operative Injection | Group C - Control
Started | 6; 7 Eyes | 7; 7 Eyes | 6; 6 Eyes
Completed | 2; 3 Eyes | 1; 1 Eyes | 2; 2 Eyes
Not Completed | 4; 4 Eyes | 6; 6 Eyes | 4; 4 Eyes
Not completed — Lost to Follow-up | 3 | 6 | 2
Not completed — Surgery cancelled | 1 | 0 | 1
Not completed — Insurance changed, standard of care visit not covered | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Not different from the assignment in Participation Flow. Participants can enroll two eyes in the study if both are eligible and trabeculectomy is recommended by the physician
Units Other Than Participants: eyes
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A - Pre-operative Injection | Group B - Intra-operative Injection | Group C - Control | Total
Number analyzed (Participants) | 6 | 7 | 6 | 19
Number analyzed (eyes) | 7 | 7 | 6 | 20
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 72.60 [68.64 to 78.17] | 72.42 [63.55 to 77.58] | 72.79 [64.72 to 79.58] | 72.60 [65.71 to 79.56]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 4 | 11
  Male | 3 | 3 | 2 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 6 | 7 | 5 | 18
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 2 | 3
  White | 5 | 5 | 2 | 12
  More than one race | 0 | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 7 | 6 | 19
Eye laterality [Count of Units; unit: eyes]
  Right eye | 3 | 4 | 3 | 10
  Left eye | 4 | 3 | 3 | 10

OUTCOME MEASURES:

1. Primary Outcome: IOP - 1 Day Postop
Description: Mean IOP at 1 day post-operatively
Time Frame: 1 day
Population: All patients who had surgery and post-operative visits were included in analysis
Measure: Mean (Standard Deviation); unit: mm Hg
Units Other Than Participants: eyes
Arm/Group | Group A - Pre-operative Injection | Group B - Intra-operative Injection | Group C - Control
Number analyzed (Participants) | 4 | 6 | 4
Number analyzed (eyes) | 5 | 6 | 4
mm Hg | 11.06 (6.60) | 10.93 (6.47) | 10.72 (6.62)
Statistical Analysis 1: Comparison: Group A - Pre-operative Injection vs Group B - Intra-operative Injection vs Group C - Control; Test type: Equivalence — ANOVA was used to analyze equivalence between arms; p = 0.52, ANOVA

2. Primary Outcome: IOP - 1 Week Postop
Description: Mean IOP at 1 week postop
Time Frame: 1 week
Population: All patients who completed postop visit were included in analysis
Measure: Mean (Standard Deviation); unit: mm Hg
Units Other Than Participants: eyes
Arm/Group | Group A - Pre-operative Injection | Group B - Intra-operative Injection | Group C - Control
Number analyzed (Participants) | 4 | 4 | 5
Number analyzed (eyes) | 5 | 4 | 5
mm Hg | 11.20 (4.49) | 9.13 (4.13) | 24.1 (8.11)
Statistical Analysis 1: Comparison: Group A - Pre-operative Injection vs Group B - Intra-operative Injection vs Group C - Control; Test type: Equivalence — Equivalence calculated using ANOVA; p = 0.01, ANOVA

3. Primary Outcome: IOP - 1 Month Postop
Description: Mean IOP 1 month postoperatively
Time Frame: 1 month
Population: All patients who completed postop visit were included in analysis
Measure: Mean (Standard Deviation); unit: mm Hg
Units Other Than Participants: eyes
Arm/Group | Group A - Pre-operative Injection | Group B - Intra-operative Injection | Group C - Control
Number analyzed (Participants) | 4 | 6 | 5
Number analyzed (eyes) | 5 | 6 | 5
mm Hg | 9.70 (3.46) | 9.67 (1.40) | 12.30 (3.23)
Statistical Analysis 1: Comparison: Group A - Pre-operative Injection vs Group B - Intra-operative Injection vs Group C - Control; Test type: Equivalence — Equivalence was assessed using ANOVA; p = 0.25, ANOVA

4. Primary Outcome: IOP - 3 Months Postop
Description: Mean IOP 3 months postoperatively
Time Frame: 3 months
Population: All patients who completed postoperative visit were included in analysis
Measure: Mean (Standard Deviation); unit: mm Hg
Units Other Than Participants: eyes
Arm/Group | Group A - Pre-operative Injection | Group B - Intra-operative Injection | Group C - Control
Number analyzed (Participants) | 4 | 4 | 5
Number analyzed (eyes) | 5 | 4 | 5
mm Hg | 11.40 (6.68) | 11.75 (1.85) | 10.6 (4.03)
Statistical Analysis 1: Comparison: Group A - Pre-operative Injection vs Group B - Intra-operative Injection vs Group C - Control; Test type: Equivalence — Equivalence determined by ANOVA; p = 0.93, ANOVA

5. Primary Outcome: IOP - 6 Months Postop
Description: Mean IOP 6 months postoperatively
Time Frame: 6 months
Population: All patients who completed postop visit were included in analysis
Measure: Mean (Standard Deviation); unit: mm Hg
Units Other Than Participants: eyes
Arm/Group | Group A - Pre-operative Injection | Group B - Intra-operative Injection | Group C - Control
Number analyzed (Participants) | 2 | 2 | 3
Number analyzed (eyes) | 3 | 2 | 3
mm Hg | 13.33 (4.62) | 12 (0) | 11.67 (2.84)
Statistical Analysis 1: Comparison: Group A - Pre-operative Injection vs Group B - Intra-operative Injection vs Group C - Control; Test type: Equivalence — Equivalence determined by ANOVA; p = 0.83, ANOVA

6. Primary Outcome: IOP - 12 Months Postop
Description: Mean IOP 12 months postoperatively
Time Frame: 12 months
Population: All participants who completed visit were included in analysis
Measure: Mean (Standard Deviation); unit: mm Hg
Units Other Than Participants: eyes
Arm/Group | Group A - Pre-operative Injection | Group B - Intra-operative Injection | Group C - Control
Number analyzed (Participants) | 2 | 1 | 2
Number analyzed (eyes) | 3 | 1 | 2
mm Hg | 14.0 (6) | 8 (NA) — cannot calculate SD with only 1 value | 10 (0)
Statistical Analysis 1: Comparison: Group A - Pre-operative Injection vs Group B - Intra-operative Injection vs Group C - Control; Test type: Equivalence — Equivalence was determined using ANOVA; p = 0.54, ANOVA

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Group A - Pre-operative Injection | Group B - Intra-operative Injection | Group C - Control
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/7 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 1/7 | 1/6
Other Adverse Events (participants affected / at risk) | 3/6 | 5/7 | 3/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A - Pre-operative Injection (N=6) | Group B - Intra-operative Injection (N=7) | Group C - Control (N=6)
Lower GI Bleed (Gastrointestinal disorders) | 0 | 0 | 1 (1)
Acute decompensated heart failure (Cardiac disorders) | 0 | 1 (1) | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A - Pre-operative Injection (N=6) | Group B - Intra-operative Injection (N=7) | Group C - Control (N=6)
Elevated intraocular pressure (IOP) (Eye disorders) | 2 (5) | 4 (6) | 3 (8)
Hyphema (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Bleb leak (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Hypotony (Eye disorders) | 0 | 2 (2) | 0
Encapsulated bleb (Eye disorders) | 0 | 1 (2) | 0 (0)
Trace anterior chamber flare (Eye disorders) | 1 (1) | 0 | 0
Ocular pain (Eye disorders) | 1 (1) | 0 | 0
Subconjunctival hemorrhage (Eye disorders) | 1 (1) | 0 | 0
Disc hemorrhage (Eye disorders) | 0 | 2 (2) | 0
Bleb dysthesia (Eye disorders) | 0 | 1 (1) | 0
Cataract progression (Eye disorders) | 0 (0) | 1 (1) | 1 (1)
Choroidal hemorrhage (Eye disorders) | 0 | 1 | 0
Retinal detachment (Eye disorders) | 0 | 1 (1) | 0

LIMITATIONS AND CAVEATS:
COVID-19 pandemic occurred during study meaning high rates of patients lost to follow-up, as non-emergent visits were canceled or postponed. This led to early termination which means we had a small number of subjects to analyze, especially those who completed all 12 months of follow-up. By the time pandemic restrictions eased, several other studies had published results on similar trials, making further enrollment unnecessary and further supporting early termination of the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-01-19): https://cdn.clinicaltrials.gov/large-docs/11/NCT03875911/Prot_SAP_002.pdf
  • Informed Consent Form (2019-04-11): https://cdn.clinicaltrials.gov/large-docs/11/NCT03875911/ICF_003.pdf